CLINICAL TRIAL: NCT00674011
Title: A Pilot Study of Hypertension in Breast Cancer Patients Receiving Bevacizumab
Brief Title: Hypertension in Breast Cancer Patients Receiving Bevacizumab
Status: Terminated | Type: Observational
Why Stopped: Slow accrual
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Erica Mayer, MD, MPH, Principal Investigator, Dana-Farber Cancer Institute
Other Study IDs: 07-149
Record Dates: First submitted 2008-05-06; First posted 2008-05-07 (Estimated); Last update posted 2014-05-06 (Estimated); Status verified 2014-05

CONDITIONS: Breast Cancer
Keywords: hypertension; bevacizumab; metastatic breast cancer
MeSH Terms: conditions — Breast Neoplasms; Hypertension | interventions — Bevacizumab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Bevacizumab — Given as part of standard of care or another research protocol

SUMMARY:
This research study will look at the effect of an anti-angiogenesis medication called Bevacizumab on blood vessels. Anti-angiogenesis medicines fight cancer by cutting off a tumor's blood supply, starving the tumor of nutrients and oxygen. Previous studies have shown these types of drugs can cause hypertension. The purpose of this study is to help researchers better understand why these drugs cause hypertension. This information will assist researchers in learning how to control this side effect.

DETAILED DESCRIPTION:
* Participants will begin this research study within 14 days of starting Bevacizumab, either as part of standard treatment or as part of another clinical trial.
* Participants will have an ultrasound test done at baseline, and after completion of their first and second cycles of therapy.
* Vital signs and blood tests will be performed a the start of the study, and after completion of the first and second cycles of therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed breast cancer
* Must be starting combination treatment with bevacizumab and chemotherapy. Treatment may not have already started. Patients may receive therapy either on or off of a clinical trial.
* Any number of prior chemotherapy or biological therapy regimens is acceptable.
* Either no history of hypertension, defined as Blood Pressure <140/90mm Hg on no antihypertensive therapy, or medically controlled pre-existing hypertension, defined as Blood Pressure < 140/90mm HG on one non-angiotensin converting enzyme inhibitor (ACE-I) or non-angiotensin receptor blocking (ARB) medication.

Exclusion Criteria:

* History of uncontrolled hypertension within the previous 6 months
* Inability to assess blood pressure or have prolonged blood pressure cuff inflation due to history of bilateral lymph node dissections, presence of an indwelling venous access device, or other condition
* Concurrent use of a statin medication
* Systolic blood pressure < 100mm Hg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with histologically or cytologically confirmed breast cancer who will be starting treatment with bevacizumab and chemotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2008-01; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
To evaluate changes in flow-mediated vasodilation (FMD) from baseline to treatment timepoints in an effort to explore the relationships between exposure to bevacizumab, eNOS activity, and vascular dysfunction. | 1 year

SECONDARY OUTCOMES:
To explore whether the development of hypertension during bevacizumab therapy correlates with vascular function | 1 year
To explore whether baseline measurements of FMD and NT are associated with the development of hypertension during bevacizumab therapy. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Erica Mayer, MD MPH, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States